CLINICAL TRIAL: NCT00439933
Title: Weight Loss in Obese Children and Adolescents and Its Effect on Improvement of Endothelial Dysfunction
Brief Title: Weight Loss in Obese Children and Adolescents and Its Effect on Improvement of Destructive Changes in Blood Vessels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1-Tafel
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2007-05-09 (Estimated); Status verified 2007-03

CONDITIONS: Obesity
Keywords: Obesity; Children; Weight loss; Endothelial dysfunction; Intervention
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Diet, Fat-Restricted

INTERVENTIONS:
Behavioral: low fat and polysaccharide rich diet
Behavioral: specific physical training program for obese children

SUMMARY:
Obesity in children and adolescents is associated with morphologic and functional changes of the vascular wall, suggesting a potential role of juvenile obesity for the development of atherosclerosis later in life. However, no evidence from intervention studies has been provided so far that weight loss in obese children can improve vascular function. Therefore we designed this study including a cohort of obese children before and after a structured weight reduction program in order to answer the question, whether such an intervention can improve vascular function and reverse destructive vascular changes.

DETAILED DESCRIPTION:
Obesity is an epidemic disease with a rapid increase in children and adolescents. According to the National Health and Nutrition Examination Surveys, the prevalence of overweight children doubled between 1976-1980 and 1999-2002 and affected 15 percent of children and adolescents in the United States. Further investigations have shown that obese children and adolescents have a high risk for the persistence of overweight into adulthood, and that morbidity and mortality are higher in those obese adults who became overweight during childhood, compared to those whose weight-gain evolved later in life. A tremendous increase in obesity-related morbidity and furthermore an immense rise in the medical costs associated with it, is to be expected. Growing evidence suggests that obesity in childhood is not only associated with a markedly increased prevalence of prediabetes or diabetes mellitus, dyslipidemia and other cardiovascular risk factors, but also predicts the development of coronary artery disease and other atherosclerotic complications in adulthood. A 55-year follow-up study showed that overweight in adolescence lead to an increased risk of morbidity and mortality from cardiovascular events. This effect is even independent of adult weight. There is evidence, that markers of early yet reversible states of atherosclerosis, such as decreased flow-mediated dilation of the brachial artery (FMD) and increased intima media thickness (IMT), correlate with measures of body weight and are predictive of cardiovascular disease.

While several studies have demonstrated that weight loss can improve metabolic risk factors in obese children, data regarding the effect on early vascular disease is missing. Therefore we designed this study including a cohort of obese children before and after a structured weight reduction program in order to answer the question, whether such an intervention can improve endothelial cell function and reverse an increased intima media thickness. Since each intervention program leading to body weight reduction is a severe interference with personal lifestyle, we feel that these questions need to be answered before intervention programs are initiated on a public health basis.

ELIGIBILITY:
Inclusion Criteria:

* children between 7 and 10 years with tanner 0 or 13 to 17 years with tanner 4 or 5
* body mass index > 97th percentile

Exclusion Criteria:

* severe medical disorders in addition to obesity
* severe psychosocial impairments
* known endocrine or genetic causes for obesity
* family history of premature cardiovascular disease
* factors affecting vascular function, including cigarette smoking
* regular medication for other diseases including vitamin supplements

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2007-04

PRIMARY OUTCOMES:
changes in flow-mediated dilation of the brachial artery
intima media thickness of the brachial artery

SECONDARY OUTCOMES:
weight reduction

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Tafel, Dr, Principal Investigator — University Hospital Heidelberg, Department of Internal Medicine I; Peter P Nawroth, Prof, Study Chair — University Hospital Heidelberg, Department of Internal Medicine I
Locations (1):
- University Hospital Heidelberg, Department of Internal Medicine I, Heidelberg, Germany